CLINICAL TRIAL: NCT00526461
Title: A Phase I Study Light Dose for Photodynamic Therapy (PDT) Using 2-[1-hexyloxyethyl]-2 Devinyl Pyropheophorbide-a (HPPH) for Treatment of Non-Small Cell Carcinoma in Situ or Non-Small Cell Microinvasive Bronchogenic Carcinoma: A Dose Ranging Study
Brief Title: Photodynamic Therapy Using HPPH in Treating Patients With Stage 0 Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000563238; RPCI-I-05903
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer
Keywords: stage 0 non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PDT using HPPH (Experimental): Patients receive HPPH IV over 1 hour on day 1. Patients then receive photodynamic therapy with laser light on day 3. Patients also undergo therapeutic bronchoscopy for endoscopic debridement on day 5.
  Interventions: Drug: HPPH

INTERVENTIONS:
Drug: HPPH — IV

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as HPPH, that is absorbed by tumor cells. The drug becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed.

PURPOSE: This phase I trial is studying the side effects and best dose of photodynamic therapy using HPPH in treating patients with stage 0 non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximally tolerated light dose (MTID) in patients with bronchogenic carcinoma in situ (CIS) or bronchogenic microinvasive carcinoma.
* To identify the systemic and normal tissue toxicity resulting from photodynamic therapy using HPPH in these patients.

Secondary

* To study tumor response in these patients.

OUTLINE: Patients receive HPPH IV over 1 hour on day 1. Approximately 2 days later, patients undergo photodynamic therapy (PDT) using laser light passed through the biopsy channel of an endoscope. Patients undergo endoscopic debridement on day 5. If viable tumor is found outside of the initial treatment area, patients may receive another dose of laser light without additional HPPH at that time.

After completion of study treatment, patients are followed at 4-6 weeks, 6 months, and periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed carcinoma in situ (CIS) or microinvasive bronchogenic non-small cell lung carcinoma

  * May have squamous cell carcinoma, adenocarcinoma, or large cell carcinoma histology
* Stage 0 (CIS or microinvasive) disease, meeting all of the following criteria:

  * Lesion must be radiographically occult and not definable by conventional CT scan of the chest
  * Lesion may or may not be invisible on white light bronchoscopy, but is definable and photographable on laser-induced fluorescence emission (LIFE) bronchoscopy
  * Biopsy of the lesion must indicate no evidence of invasion beyond cartilage on histopathology, but may be invasive through the basement membrane (microinvasive carcinoma)
* No evidence of major pulmonary vessel encasement on CT scan of the chest

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% OR ECOG PS 0-2
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 4,000/mm^3
* Prothrombin time ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 3.0 mg/dL
* Creatinine ≤ 3.0 mg/dL
* Alkaline phosphatase (hepatic) or SGOT ≤ 3 times ULN
* No porphyria or hypersensitivity to porphyrin or porphyrin-like compounds
* No severe chronic obstructive pulmonary disease, that in the opinion of the investigator, would preclude multiple bronchoscopies or partial central airway obstruction from mucous/debris formation
* Patients with underlying lung disease must be judged (by the principal investigator) able to withstand mucous or debris formation at the site of treatment
* No contraindications for bronchoscopy
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior and no concurrent chemotherapy or radiotherapy
* Prior therapy of any type (e.g., chemotherapy or radiotherapy) allowed for lung cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-02; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Toxicity as measured by NCI CTC v2.0 | Daily while in-house, weekly after discharge, at 4-6 weeks and at 6 months

SECONDARY OUTCOMES:
Tumor response | At 4-6 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samjot Dhillon, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States